CLINICAL TRIAL: NCT05857969
Title: Adopting a Functional Precision Medicine Approach For Individualized Pediatric Cancer Treatments
Brief Title: Ex Vivo Drug Sensitivity Testing and Multi-Omics Profiling
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other); First Ascent Biomedical Inc. (Industry); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Diana Azzam, PhD, Assistant Professor, Florida International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112215; 2U54MD012393-06 (NIH)
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Large Cell Lymphoma; Refractory Childhood Acute Lymphoblastic Leukemia; Refractory Childhood Hodgkin Lymphoma; Refractory Childhood Malignant Germ Cell Neoplasm; Recurrent Childhood Brain Tumor; Recurrent Childhood Brainstem Glioma; Recurrent Childhood Rhabdomyosarcoma; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Childhood Ependymoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Gliosarcoma; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Childhood Malignant Solid Neoplasm; Recurrent Childhood Malignant Solid Neoplasm; Recurrent Childhood Malignant Neoplasm; Refractory Childhood Malignant Neoplasm
Keywords: ex vivo drug sensitivity assay; genomic profiling; Functional precision medicine; Biomarker development
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Familial ependymoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Functional Precision Medicine for Chemorefractory or relapsed patients (Experimental): We intend to enroll chemorefractory or relapsed pediatric patients with all types of cancers where tumor tissue would be available for functional precision medicine that integrates ex vivo drug screening and genomic profiling. The results of the drug sensitivity assay and genetic screening will be used to inform treating physician about patient-specific drug sensitivity or resistance guiding best therapy choices.
  Interventions: Device: Functional Precision Medicine

INTERVENTIONS:
Device: Functional Precision Medicine — Ex Vivo Drug Sensitivity Testing + Genomic Tumor Profiling

SUMMARY:
Functional precision medicine (FPM) is a relatively new approach to cancer therapy based on direct exposure of patient- isolated tumor cells to clinically approved drugs and integrates ex vivo drug sensitivity testing (DST) and genomic profiling to determine the optimal individualized therapy for cancer patients. In this study, we will enroll relapsed or refractory pediatric cancer patients with tissue available for DST and genomic profiling from the South Florida area, which is 69% Hispanic and 18% Black. Tumor cells collected from tissue taken during routine biopsy or surgery will be tested.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: The primary objective of the study is to determine feasibility of providing pediatric cancer patients with access to personalized treatment options and clinical management recommendations based on Functional Precision Medicine (FPM), the combination of ex vivo drug sensitivity testing (DST) and genomic profiling.

SECONDARY OBJECTIVE: The secondary objective of the study is to compare individual outcomes (response and disease-free survival) in patients with pediatric cancers treated with FPM-guided therapy as compared to non-FPM guided (conventional) therapy.

EXPLORATORY OBJECTIVE: To explore associations between tumor molecular characteristics (genomic and transcriptomic variation) and ex vivo drug response with respect to patient ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 years or younger at the time of enrollment on this study of any gender, race or ethnicity.

Subjects with suspected or confirmed diagnosis of recurrent or refractory cancer Subjects who are scheduled for or have recently had biopsy or tumor excised (solid tumors) or bone marrow aspirate (blood cancers) Subjects willing to have a blood draw or buccal swab done for the purposes of genetic testing Subjects or their parents or legal guardians willing to sign informed consent Subjects aged 7 to 17 willing to sign assent

Exclusion Criteria:

* Subjects who do not have malignant tissue available and accessible The amount of excised malignant tissue is not sufficient for the ex vivo drug testing and/or genetic profiling.

Patients with newly diagnosed tumors and tumors that have high (>90%) cure rate with safe standard therapy.

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2028-02-22 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients that receive Functional Precision Medicine (FPM)-guided treatment options | Up to 6 years
  This study will be considered successful (feasibility demonstrated) if it is possible to choose and initiate a monotherapy or combination drug regimen based on functional and/or genomics data within 4 weeks in at least 39 out of 65 patients (60%).
  To achieve at least 90% power, the null hypothesis will be rejected when at least 39 out of 65 patients receive treatment recommendations through functional and/or genomics data within 4 weeks on the study.
  With that outcome, we would have 95% confidence that the true feasibility rate is at least 40% (95% CI: 0.4905 to 1).

SECONDARY OUTCOMES:
Assessing Progression-Free Survival (PFS) in FPM-guided therapy versus standard of care | Up to 6 years
  We will assess changes in cohort PFS by comparing PFS in patients treated with FPM-guided therapy versus PFS in patients treated with non-FPM guided conventional therapy (standard of care)
Assessing Previous vs Trial PFS Ratio (PFS2/PFS1) in FPM-guided patients versus standard of care | Up to 6 years
  We will assess changes in PFS from each patient's previous treatment versus their PFS from the treatment assigned during the trial. Assessments will be made both in the FPM-guided cohort and the non-FPM-guided cohort (standard of care). Analysis will include both the raw ratio as well as the number of incidences of 30% improved PFS on trial versus previous regimen (PFS2/PFS1 > 1.3x).
Assessing Overall Survival (OS) in FPM-guided patients versus standard of care patients | Up to 6 years
  We will assess changes in cohort OS by comparing OS in patients treated with FPM-guided therapy versus OS in patients treated with non-FPM guided conventional therapy (standard of care)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Azzam, Principal Investigator — Florida International University; Maggie Fader, Principal Investigator — Nicklaus Children's Hospital
Locations (1):
- Nicklaus Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No